CLINICAL TRIAL: NCT04183946
Title: Willkommen Mutterglück: A Controlled Trial of Internet Based Cognitive Behavioural Therapy (CBT) for Pregnant and Postpartum Women With Depression and Anxiety
Brief Title: Willkommen Mutterglück: Online CBT for Pregnant and Postpartum Women With Depression and Anxiety
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: University of Zurich (Other)
Collaborators: Ambulatorium für kognitive Verhaltenstherapie und Verhaltensmedizin - UZH (Unknown); Lamprecht AG (Unknown)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: Willkommen Mutterglück Program
Record Dates: First submitted 2018-04-11; First posted 2019-12-03 (Actual); Last update posted 2019-12-03 (Actual); Status verified 2019-11

CONDITIONS: Prenatal Anxiety; Generalized Anxiety; Postpartum Depression; Major Depressive Disorder
Keywords: generalized anxiety disorder; depression; cognitive behavioral therapy; web-based cognitive behavioural therapy; web-based CBT; pregnancy; prenatal depression; prenatal anxiety; postpartum anxiety; postpartum depression
MeSH Terms: conditions — Generalized Anxiety Disorder; Depression, Postpartum; Depressive Disorder, Major; Depression

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Online Cognitive Behavioural Therapy (Other): Screened participants diagnosed with minor to moderate anxiety and/or depression will receive online CBT therapy (8 interactive sessions) aiming to treat their symptomatology. Each session can be completed at one's own pace.
  Interventions: Behavioral: Online Cognitive Behavioural Therapy

INTERVENTIONS:
Behavioral: Online Cognitive Behavioural Therapy — The "Willkommen Mutterglück" program is an 8-session, interactive web-based CBT intervention for prenatal and postpartum depression and anxiety. The sessions are administered online via audio and video images. Each weekly session has a duration of 40-50 minutes during which the participants are asked to actively participate through exercises and quizzes.
  A SCID interview for screening will be conducted by a trained clinical psychologist and an experienced psychiatrist from our outpatient clinic will verify the diagnosis. Screened and consented participants will answer baseline questionnaires, provide sociodemographic information and receive a private login to access the program. After completing the 2nd, 4th and 8th intervention session participants will fill in psychological questionnaires.
  During the intervention, participants will be contacted three times by telephone by coaches (psychotherapists in training) who follow a manualized script.
  Other Names: Willkommen Mutterglück: Online CBT program for pre-postnatal depression & anxiety

SUMMARY:
This intervention study aims to evaluate the effectivity of web-based cognitive therapy in reducing depression and anxiety in pregnant and postpartum women. Moreover, it aims to assess treatment feasibility and usability of the treatment in the same population.

After an initial screening to determine the eligibility to participate, all participants fulfilling the inclusion criteria will receive their personal access login in order to start the intervention.

DETAILED DESCRIPTION:
Introduction: Evidence has shown that 10-20% of women suffer from depression during gestation and after birth (Barnes, 2014; Zaers, Waschke & Ehlert, 2008), while 7-21% present clinically relevant anxiety levels prenatally and following delivery (Grant, McMahon & Austin, 2008).

Previous research has shown that if a woman has high levels of depression or anxiety during pregnancy her child is at about double the risk for attention deficit hyperactivity disorder, conduct disorders, difficult temperament and behavioural problems later in development (O'Connor et al., 2002). High levels of prenatal anxiety and depression are frequently comorbid (Amiel Castro et al., 2016) and together with stress have been shown to increase risk for preterm delivery, low birth weight, impaired memory and cognitive function among others (Talge, Neal & Glover, 2007). The important biopsychological changes brought by the perinatal period (Ehlert et al., 1990) require constant attention from health workers since they carry relevant risk factors for the mother's health and for the infant's neurodevelopment (Schetter & Tanner, 2012).

Current depression interventions are not deliverable to a large number of individuals (Andersson & Titov, 2014). As seen worldwide, the difficulty to receive proper treatment for depression and anxiety is also evident in Switzerland. About half of people suffering from depression and/or anxiety are not diagnosed and consequently do not receive any sort of psychological or pharmaceutical treatment (Baer et al., 2013).

The internet offers an opportunity to deliver tailored interventions such as those based on cognitive behavioural therapy (CBT) to a large audience, cost-effectively, while preserving intervention fidelity and anonymity. The potential effectiveness of the internet is indicated by research demonstrating the successful delivery of CBT by computer and the use of the internet in the delivery of CBT treatment (Andrews et al., 2010). Recent reviews of the evidence have recommended further research that includes long-term follow-up and evaluation of novel treatment modalities such as the ones provided by internet (Dennis et al., 2012). Moreover, online interventions have been widely explored for different mental health problems (Sourander et al., 2016) suggesting its potential to increase access to and uptake of services for women with a perinatal disorder.

The "Willkommen Mutterglück" program is an 8-session, interactive web-based cognitive behavioural intervention for prenatal and postpartum depression and anxiety.

Given the prevalence rates of depression and anxiety during the perinatal period and the rates of untreated patients, it is important to propose treatment alternatives. Several reviews on the area emphasize that topics such as type and amount of CBT material incorporated to the program, length and frequency of sessions, amount of homework given and frequency of minimal therapist intervention are related to effectivity of online interventions and warrant further research. Also, it is unclear whether therapist contact focusing on motivation to complete the program is more effective than non-therapist contact in the treatment of the disorders. Therefore, routine use of this online intervention for depressed and anxious mothers is only possible if this program/the effects are is scientifically evaluated with biomarkers.

The primary goal of this project is to investigate the effectiveness of an online cognitive behavioural intervention specifically tailored to pregnant and postpartum women in reducing depression and anxiety symptoms. The secondary goal is to assess the feasibility and usability of this intervention on the treatment of depression and anxiety.

Method: The investigators aim to recruit N=300 patients from the first gestational trimester to one year after birth. The eight intervention sessions are administered online via audio and video images. The participants are asked to actively participate during their weekly session through exercises and quizzes. Each weekly session has a duration of 40-50 minutes.

A SCID interview for screening will be conducted by a trained clinical psychologist and an experienced psychiatrist from a trusted Outpatient Clinic will verify the diagnosis. Screened and consented participants will then fill in some baseline questionnaires, provide sociodemographic information and receive a private login to access the program in order to start the intervention. After completing the second, fourth and eight intervention session participants will fill in the same and other psychological questionnaires.

Throughout the intervention, the investigators will frequently monitor patient's progress and potential worsening of depressive and anxiety symptoms. The investigating team will be particularly attentive to suicidal ideation. Patients identified with suicidal thoughts will be immediately contacted by the study team and advised to an appropriate course of action. Moreover, in all online pages of the "Willkommen Mutterglück" intervention participants can find an SOS button, providing contact information of emergency psychiatric units and suicide hotlines.

During the online intervention, participants will be contacted three times by telephone by coaches (psychotherapists in training). The content of coaching calls will adhere to a manualized script with defined aims of reviewing patient's progress, problem solving, encourage skill acquisition and introducing topics in upcoming sessions. Coaches will be trained with a specific manual developed by the investigation team. Training for the coaching role will involve reading the coach manual, knowledge of the program content and explanations from a senior researcher about the role and the tasks involved.

Importance: In view of the substantial challenge posed by the global burden of depression and anxiety, it is relevant to investigate how a disorder, which is a leading cause of disability worldwide, may affect mothers and mothers-to-be. Pregnant and postpartum women are often reluctant to take medication due to concerns about breast milk transmission or potential side effects. Therefore, non-pharmacologic interventions are a desirable first-line treatment option for this population. Given that despite frequent interactions with health workers during pregnancy and postpartum, rates of treatment for perinatal disorders are low, online therapy may be a viable treatment alternative. The planned longitudinal study is relevant in investigating the feasibility of an interactive CBT online intervention including minimal psychotherapist involvement and tailored specifically for this population. At the same time, it assesses the effectiveness of it in reducing depression and/or anxiety in pregnant and postpartum women. The results will help to better understand if an intervention (online program with coaching) with few barriers (e.g. no travel, no childcare costs, reduced stigma), may serve as an effective treatment option for pregnant and postpartum women who experience significant stigma or are underresourced in their local community.

ELIGIBILITY:
Inclusion Criteria:

* pregnant women or women who had given birth in the last year
* between 18 and 45 years old
* minor to moderate depression and/or generalised anxiety disorder
* fluent in German
* having a computer, laptop or handheld device with internet access

Exclusion Criteria:

* women with a severe medical disorder or a severe psychological disorder such as psychosis, drug addiction and other substance abuse
* women taking psychotropic medication
* women with current suicidality
* women who are currently receiving psychological treatment for depression or anxiety

Ages: 18 Years to 45 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 300 (Estimated)
Dates: Start 2020-06 (Estimated); Primary Completion 2022-01 (Estimated); Study Completion 2024-01 (Estimated)

PRIMARY OUTCOMES:
Change of depressive symptoms at four measuring points from baseline to follow up | At baseline, during week 4, 8, 16 of the intervention and at one month after completing intervention.
  Measured with Beck's Depression Inventory (BDI)
Change of anxiety symptoms at four measuring points from baseline to follow up | At baseline, during week 4, 8, 16 of the intervention and at one month after completing intervention.
  Measured with Beck's Anxiety Inventory (BAI)
Change of severity of depressive symptoms at four measuring points from baseline to follow up | At baseline, during week 4, 8, 16 of the intervention and at one month after completing intervention.
  Measured with Patient Health Questionnaire (PHQ) Ranges from 0-27 (0-4=none-minimal; 5-9=mild; 10-14=moderate; 15-19=moderately severe; 20-27=severe)
Change of depression symptoms from baseline until follow-up | At baseline and during week 16 of the intervention
  Measured with Edinburgh Postnatal Depression Scale (EPDS) Minimum score = 0, maximum score = 30. Cut off value is set at 12/13

SECONDARY OUTCOMES:
Participant's satisfaction with the program and it's usability | At week 16 of the intervention
  This is reported with open-ended questions about satisfaction with the program and with self-report measure that assesses the patient's attitude on the overall usability to the program (System Usability Scale, SUS) The scores range from 0-100. It is agreed that score above 68 would be considered above average, whilst scores below 68 would be considered below average.
Program's evaluation of feasibility with prenatal and postpartum women | From baseline until 1 month follow-up of the intervention
  This is reported with user engagement, such as duration spent on web-intervention-site and number of log-ins into the intervention. These different measures should give an overview over how the participants perceive and evaluate the program and how they rate its feasibility.

CONTACTS AND LOCATIONS:
Overall Officials: Ulrike Ehlert, Prof. Dr., Study Chair — University of Zurich, Department of Psychology - Clinical Psychology and Psychotherapy; Rita Amiel Castro, Dr. phil., Principal Investigator — University of Zurich, Department of Psychology - Clinical Psychology and Psychotherapy
Locations (1):
- University of Zurich, Department of Psychology - Clinical Psychology and Psychotherapy, Zurich, Switzerland

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Background] Amiel Castro RT, Pinard Anderman C, Glover V, O'Connor TG, Ehlert U, Kammerer M. Associated symptoms of depression: patterns of change during pregnancy. Arch Womens Ment Health. 2017 Aug;20(4):593-594. doi: 10.1007/s00737-017-0728-7. Epub 2017 May 25. No abstract available. PMID 28540597
- [Background] Andersson G, Titov N. Advantages and limitations of Internet-based interventions for common mental disorders. World Psychiatry. 2014 Feb;13(1):4-11. doi: 10.1002/wps.20083. PMID 24497236
- [Background] Andrews G, Cuijpers P, Craske MG, McEvoy P, Titov N. Computer therapy for the anxiety and depressive disorders is effective, acceptable and practical health care: a meta-analysis. PLoS One. 2010 Oct 13;5(10):e13196. doi: 10.1371/journal.pone.0013196. PMID 20967242
- [Background] Barnes M, Cox J, Doyle B, Reed R. Evaluation of a practice-development initiative to improve breastfeeding rates. J Perinat Educ. 2010 Fall;19(4):17-23. doi: 10.1624/105812410X530893. PMID 21886418
- [Background] Ehlert U, Patalla U, Kirschbaum C, Piedmont E, Hellhammer DH. Postpartum blues: salivary cortisol and psychological factors. J Psychosom Res. 1990;34(3):319-25. doi: 10.1016/0022-3999(90)90088-l. PMID 2342000
- [Background] Grant KA, McMahon C, Austin MP. Maternal anxiety during the transition to parenthood: a prospective study. J Affect Disord. 2008 May;108(1-2):101-11. doi: 10.1016/j.jad.2007.10.002. Epub 2007 Nov 14. PMID 18001841
- [Background] Griffiths KM, Farrer L, Christensen H. The efficacy of internet interventions for depression and anxiety disorders: a review of randomised controlled trials. Med J Aust. 2010 Jun 7;192(S11):S4-11. doi: 10.5694/j.1326-5377.2010.tb03685.x. PMID 20528707
- [Background] Hofmann SG, Asnaani A, Vonk IJ, Sawyer AT, Fang A. The Efficacy of Cognitive Behavioral Therapy: A Review of Meta-analyses. Cognit Ther Res. 2012 Oct 1;36(5):427-440. doi: 10.1007/s10608-012-9476-1. Epub 2012 Jul 31. PMID 23459093
- [Background] O'Connor TG, Heron J, Glover V; Alspac Study Team. Antenatal anxiety predicts child behavioral/emotional problems independently of postnatal depression. J Am Acad Child Adolesc Psychiatry. 2002 Dec;41(12):1470-7. doi: 10.1097/00004583-200212000-00019. PMID 12447034
- [Background] Richards D, Richardson T. Computer-based psychological treatments for depression: a systematic review and meta-analysis. Clin Psychol Rev. 2012 Jun;32(4):329-42. doi: 10.1016/j.cpr.2012.02.004. Epub 2012 Feb 28. PMID 22466510
- [Background] Dunkel Schetter C, Tanner L. Anxiety, depression and stress in pregnancy: implications for mothers, children, research, and practice. Curr Opin Psychiatry. 2012 Mar;25(2):141-8. doi: 10.1097/YCO.0b013e3283503680. PMID 22262028
- [Background] Sourander A, McGrath PJ, Ristkari T, Cunningham C, Huttunen J, Lingley-Pottie P, Hinkka-Yli-Salomaki S, Kinnunen M, Vuorio J, Sinokki A, Fossum S, Unruh A. Internet-Assisted Parent Training Intervention for Disruptive Behavior in 4-Year-Old Children: A Randomized Clinical Trial. JAMA Psychiatry. 2016 Apr;73(4):378-87. doi: 10.1001/jamapsychiatry.2015.3411. PMID 26913614
- [Background] Talge NM, Neal C, Glover V; Early Stress, Translational Research and Prevention Science Network: Fetal and Neonatal Experience on Child and Adolescent Mental Health. Antenatal maternal stress and long-term effects on child neurodevelopment: how and why? J Child Psychol Psychiatry. 2007 Mar-Apr;48(3-4):245-61. doi: 10.1111/j.1469-7610.2006.01714.x. PMID 17355398
- [Background] Zaers S, Waschke M, Ehlert U. Depressive symptoms and symptoms of post-traumatic stress disorder in women after childbirth. J Psychosom Obstet Gynaecol. 2008 Mar;29(1):61-71. doi: 10.1080/01674820701804324. PMID 18266166
- [Background] Alder J, Urech C. Angststörungen in der Schwangerschaft. In: Riecher-Rössler A, eds. Psychische Erkrankungen in Schwangerschaft und Stillzeit. Basel, Switzerland: Karger; 2014.
- [Background] Amiel Castro R, Glover V, Kammerer M, Ehlert U. Associations between maternal symptoms of depression, coping strategies and infant temperament: A longitudinal study from pregnancy to postpartum, Manuscript submitted for publication.
- [Background] Baer N, Schuler D, Moreau-gruet F. Depressionen in der Schweizer Bevölkerung Daten zur Epidemiologie, Behandlung und sozial-beruflichen Integration. Obsan Bericht 56, 2013.
- [Background] Bergant AM, Nguyen T, Heim K, Ulmer H, Dapunt O. [German language version and validation of the Edinburgh postnatal depression scale]. Dtsch Med Wochenschr. 1998 Jan 16;123(3):35-40. doi: 10.1055/s-2007-1023895. German. PMID 9472218
- [Background] Carter D, Kostaras X. Psychiatric disorders in pregnancy. British Columbia Medical Journal 47(2): 96-100, 2005.
- [Background] Gast U, Oswald T, Zündorf F, Hofmann A. SKID-D- Strukturiertes Klinisches Interview für DSM-IV. Dissoziative Störungen Manual. Göttingen, Germany: Hogrefe; 2000.
- [Background] Hautzunger M, Keller F, Kühner C. Beck Depressions-Inventar Revision. Manual. München, Germany: Pearson; 2009.
- [Background] Löwe B, Zipfel S, Herzog W. Deutsche Übersetzung und Validierung des Brief Patient Health Questionnaire (Brief PHQ). Medizinische Universitätsklinik Heidelberg, Germany: AOK, no date.
- [Background] Margraf J, Ehlers A. Beck-Angst-Inventar. Manual. München, Germany: Pearson; 2007.
- [Background] Oates MR. Perinatal psychiatric syndromes: clinical features. Psychiatry, 5(1): 5-9, 2006.
- [Background] O'Hara MW, Swain AM. Rates and risk of postpartum depression-a meta-analysis. International Review of Psychiatry 8(1): 37-54, 1996.
- [Background] Pössel P, Seemann S, Hautzinger M. Evaluation eines deutschsprachigen Instrumentes zur Erfassung positiver und negativer automatischer Gedanken. Evaluation of a German-language instrument for assessing positive and negative automatic thoughts. Zeitschrift Für Klinische Psychologie Und Psychotherapie: Forschung Und Praxis 34(1): 27-34, 2005.
- [Background] Rummel B, Ruegenhagen E, Reinhardt W. Fragebogen zur System-Gebrauchstauglichkeit; 2013.
- See also: Pregnancy related research by the University of Zurich — http://www.ichbinschwanger.ch